CLINICAL TRIAL: NCT02653417
Title: A Randomized, Double-Blind, Placebo-Controlled, Dose Ranging Study to Evaluate the Safety and Efficacy of RAD1901 in Postmenopausal Women With Moderate to Severe Vasomotor Symptoms
Brief Title: Study to Evaluate the Safety and Efficacy of RAD1901 in Postmenopausal Women With Moderate to Severe Vasomotor Symptoms
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor's Decision
Sponsor: Radius Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VMRAD1901-203
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2019-03-13 (Actual); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Vasomotor Symptoms; Hot Flashes
MeSH Terms: conditions — Hot Flashes | interventions — RAD1901; elacestrant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen 1 (Experimental): RAD1901 5 mg/day
  Interventions: Drug: RAD1901
- Regimen 2 (Experimental): RAD1901 10 mg/day
  Interventions: Drug: RAD1901
- Regimen 3 (Experimental): RAD1901 20 mg/day
  Interventions: Drug: RAD1901
- Regimen 4 (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: RAD1901 — RAD1901
  Other Names: Elacestrant
  Arms: Regimen 1; Regimen 2; Regimen 3
Other: Placebo — Placebo
  Arms: Regimen 4

SUMMARY:
The primary objective of this study was to determine the clinical safety of RAD1901 and to evaluate whether RAD1901 reduced the frequency and severity of moderate to severe vasomotor symptoms (VMS; "hot flashes") in postmenopausal women.

DETAILED DESCRIPTION:
This was a Phase 2b outpatient, prospective, multicenter, double-blind, randomized, placebo-controlled study to determine whether elacestrant reduces the frequency and severity of vasomotor symptoms (VMS; "hot flashes") in postmenopausal women with moderate to severe hot flashes. Postmenopausal women who met study criteria were followed for 12 weeks on double-blind study medication and two weeks off study medication.

Treatment was randomized 1:1:1:1 to ensure that an approximately equal number of patients were exposed to each of three RAD1901 (elacestrant) doses (5, 10 and 20 mg/day) or placebo. The total period of placebo exposure was 14 weeks.

Enrolling approximately 300 patients was expected to provide power for testing superiority of the primary efficacy endpoint outcomes.

ELIGIBILITY:
Inclusion Criteria:

To have participated in this study, a subject MUST:

1. be a postmenopausal woman between 40 and 65 years of age, inclusive
2. be seeking relief or treatment for moderate to severe VMS
3. be willing to discontinue and abstain from the following: vaginal hormonal products; transdermal or oral estrogen or estrogen/progestin combination; progestin implants; injectable estrogen; topical progesterone cream, selective estrogen receptor modulators and intrauterine devices (IUDs)
4. have no clinically significant abnormalities on pelvic exam except for vulvovaginal atrophy (VVA)
5. have a normal or clinically insignificant transvaginal ultrasound (TVU) with an endometrial thickness <4 mm at screening
6. have a normal endometrial biopsy subsequent to the TVU without clinically relevant results
7. have a normal screening Papanicolaou (Pap) smear
8. have a mammogram within 9 months prior to randomization. Subjects must have had a Breast Imaging Reporting and Data System (BI-RADS) mammography result of 1 or 2 to enroll.

Exclusion Criteria:

Subjects with any of the following characteristics were not be eligible to participate in the study:

1. have a history of invasive breast cancer or ductal carcinoma in situ, melanoma or any gynecologic cancer.
2. using any of the following:

   * oral estrogen-, progestin-, androgen-, or selective estrogen receptor modulator (SERM) containing drug products within 8 weeks before screening (visit 1)
   * transdermal hormone products within 4 weeks before screening (visit 1)
   * vaginal hormone products (rings, creams, gels) within 4 weeks before screening (visit 1)
   * progestin implants/injectables, IUDs or estrogen pellets/injectables within 6 months before screening (visit 1)
   * anabolic steroids
3. have been treated with a gonadotropin-releasing hormone (GnRH) agonist within the last year
4. have been treated with anti-estrogens or aromatase inhibitors within 2 months prior to study entry
5. have been concurrently treated and will abstain from gabapentin and paroxetine or serotonin and norepinephrine reuptake inhibitors (SNRIs) for VMS or other indications for 3 months during the trial and have not taken within 4 weeks prior to screening
6. have unexplained vaginal bleeding within the 3 months prior to study entry
7. have an endometrial biopsy at baseline with a diagnosis by a gynecologic pathologist of proliferative, hyperplasia, polyp or cancer
8. have unresolved cervical cytological smear report of atypical glandular or squamous cells of undetermined significance. Cervical cytologic smear report of ASCUS, low grade squamous intraepithelial lesion or greater, or any reported dysplasia
9. have unresolved findings suspicious for malignancy on the breast examination

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 139 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12-12 (Actual); Study Completion 2018-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Radius Pharmaceuticals, Inc.
Locations (1):
- Women's Health Care Specialists P.C. - Beyer Research, Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Regimen 1: RAD1901 5 mg
  RAD1901: RAD1901
- Regimen 2: RAD1901 10 mg
  RAD1901: RAD1901
- Regimen 3: RAD1901 20 mg
  RAD1901: RAD1901
Period: Overall Study
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 | Regimen 4
Started | 38 | 34 | 29 | 38
Completed | 37 | 32 | 26 | 33
Not Completed | 1 | 2 | 3 | 5

BASELINE CHARACTERISTICS:
Population: mITT population
Groups:
- Regimen 1 RAD1901 5 mg: RAD1901 5 mg
  RAD1901: RAD1901
- Regimen 2 RAD1901 10 mg: RAD1901 10 mg
  RAD1901: RAD1901
- Regimen 3 RAD1901 20 mg: RAD1901 20 mg
  RAD1901: RAD1901
- Regimen 4 Placebo: Placebo
  Placebo: Placebo
- Total: Total of all reporting groups
Arm/Group | Regimen 1 RAD1901 5 mg | Regimen 2 RAD1901 10 mg | Regimen 3 RAD1901 20 mg | Regimen 4 Placebo | Total
Number analyzed (Participants) | 38 | 34 | 28 | 38 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (4.83) | 55.4 (5.08) | 54.1 (4.07) | 53.9 (5.09) | 55.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 34 | 28 | 38 | 138
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 8 | 7 | 6 | 29
  Not Hispanic or Latino | 30 | 26 | 21 | 32 | 109
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1 | 1 | 3
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 12 | 6 | 10 | 34
  White | 30 | 22 | 21 | 27 | 100
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 38 | 34 | 28 | 38 | 138

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in the Frequency of Moderate to Severe Hot Flashes
Description: Change from baseline to week 12 in the average number of moderate and severe hot flashes per day, where change is calculated as week 12 minus baseline so that negative values indicate a reduction (improvement) of hot flash frequency.
  Severity of hot flashes was self-assessed and reported as follows:
  * Mild: sensation of heat without sweating
  * Moderate: sensation of heat with sweating, able to continue activity
  * Severe: sensation of heat with sweating, causing cessation of activity.
Time Frame: Baseline and 12 weeks
Population: The modified intent to treat (mITT) population was used. This included all patients in the safety population who had recorded hot flash data in their eDiaries for at least 5 days during baseline and for at least one day while on double-blind study medication, and was the primary analysis population for all efficacy analyses
Measure: Least Squares Mean (Standard Error); unit: moderate to severe hot flashes per day
Arm/Group | Regimen 1 | Regimen 2 | Regimen 3 | Regimen 4
Number analyzed (Participants) | 38 | 34 | 28 | 38
moderate to severe hot flashes per day | -3.48 (0.793) | -3.74 (0.867) | -4.12 (0.944) | -3.66 (0.808)
Statistical Analysis 1: Comparison: Regimen 1 vs Regimen 4; Regimen 1 = 5 mg vs Regimen 4 = placebo; Test type: Superiority; Mean Difference (Final Values) = -0.18
Statistical Analysis 2: Comparison: Regimen 2 vs Regimen 4; Regimen 2 = 10 mg vs Regimen 4 = placebo; Test type: Superiority; Mean Difference (Final Values) = 0.08
Statistical Analysis 3: Comparison: Regimen 3 vs Regimen 4; Regimen 3 = 20 mg vs Regimen 4 = placebo; Test type: Superiority; Mean Difference (Final Values) = 0.46

2. Secondary Outcome: Change From Baseline to Week 4 in the Frequency of Moderate to Severe Hot Flashes
Description: Change from baseline to week 4 in the average number of moderate and severe hot flashes per day, where change is calculated as week 4 minus baseline so that negative values indicate a reduction (improvement) of hot flash frequency.
Time Frame: Baseline and 4 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: moderate to severe hot flashes per day
Arm/Group | Regimen 1 RAD1901 5 mg | Regimen 2 RAD1901 10 mg | Regimen 3 RAD1901 20 mg | Regimen 4 Placebo
Number analyzed (Participants) | 38 | 34 | 28 | 38
moderate to severe hot flashes per day | -1.15 (3.644) | -2.22 (4.872) | -2.70 (3.764) | -3 (4.075)

3. Secondary Outcome: Change From Baseline to Week 4 and Week 12 in the Severity of Hot Flashes
Description: Change from baseline to week 4 and week 12 in the average daily severity of hot flashes, where change is calculated as week 4 or week 12 minus baseline so that negative values indicate a reduction (improvement) of hot flash severity.
  Subjects recorded the number of hot flashes per day using an electronic diary. Daily severity score for hot flashes for each subject was calculated as the sum of the number of mild hot flashes, plus 2 times the number of moderate hot flashes, plus 3 times the number of severe hot flashes, divided by the total number of mild, moderate, and severe hot flashes. That is,
  Daily Severity Score = (Fmild + 2•Fmod + 3•Fsev)/(Fmild + Fmod + Fsev) where Fmild= frequency of mild hot flashes, Fmod = frequency of moderate hot flashes, Fsev = frequency of severe hot flashes.
  The measure is a weighted average of the frequencies of Hot Flashes.
Time Frame: Baseline, 4 weeks, and 12 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: hot flash severity score per day
Arm/Group | Regimen 1 RAD1901 5 mg | Regimen 2 RAD1901 10 mg | Regimen 3 RAD1901 20 mg | Regimen 4 Placebo
Number analyzed (Participants) | 38 | 34 | 28 | 38
hot flash severity score per day
  Week 4 change from baseline in severity | -0.04 (0.25) | -0.07 (0.26) | -0.13 (0.273) | -0.00 (0.280)
  Week 12 change from baseline in severity | -0.09 (0.337) | -0.08 (0.373) | -0.13 (0.313) | -0.01 (0.409)

4. Secondary Outcome: Change From Baseline to Week 4 and Week 12 in the Frequency of All Hot Flashes
Description: Change from baseline to week 4 and week 12 in the average number of all hot flashes (mild, moderate, and severe) by eDiary, where change is calculated as week 4 or week 12 minus baseline so that negative values indicate a reduction (improvement) of hot flash frequency.
Time Frame: Baseline, 4 weeks, and 12 weeks
Population: mITT population
Measure: Mean (Standard Deviation); unit: hot flashes per day
Arm/Group | Regimen 1 RAD1901 5 mg | Regimen 2 RAD1901 10 mg | Regimen 3 RAD1901 20 mg | Regimen 4 Placebo
Number analyzed (Participants) | 38 | 34 | 28 | 38
hot flashes per day
  Week 4 change from baseline | -0.99 (3.803) | -2.23 (4.792) | -2.29 (3.754) | -3.27 (4.107)
  Week 12 change from baseline | -3.47 (5.076) | -2.40 (3.560) | -3.91 (5.263) | -3.74 (4.228)

ADVERSE EVENTS:
Time Frame: Up to 14 weeks
Arm/Group | Regimen 1 RAD1901 5 mg | Regimen 2 RAD1901 10 mg | Regimen 3 RAD1901 20 mg | Regimen 4 Placebo
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/34 | 0/29 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/34 | 0/29 | 0/38
Other Adverse Events (participants affected / at risk) | 11/38 | 3/34 | 7/29 | 13/38
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Regimen 1 RAD1901 5 mg (N=38) | Regimen 2 RAD1901 10 mg (N=34) | Regimen 3 RAD1901 20 mg (N=29) | Regimen 4 Placebo (N=38)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 4
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 2 | 1
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 2 | 2
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 2
Vaginal haemorrhage (Reproductive system and breast disorders) | 2 | 1 | 1 | 4
Headache (Nervous system disorders) | 2 | 1 | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2
Insomnia (Psychiatric disorders) | 2 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No